CLINICAL TRIAL: NCT01100697
Title: Fetal Spina Bifida -Prenatal Course and Outcome in 103 Cases A Single Center Experience.
Brief Title: Outcome of Fetal Spina Bifida
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Daniel Alexander Beyer, Dr. D. A. Beyer, University of Luebeck
Other Study IDs: UKSH-HL-09-181
Record Dates: First submitted 2010-04-02; First posted 2010-04-09 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy; Fetal and Neonatal Health
Keywords: prenatal diagnosis; ultrasound; outcome; spina bifida; neural tube defect
MeSH Terms: conditions — Spinal Dysraphism; Neural Tube Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- thoracal lesion: spinal lesion at thoracal level detected at prenatal ultrasound exam
- lumbar lesion: spinal lesion at lumbar level detected at prenatal ultrasound exam
- sacral lesion: spinal lesion at sacral level detected at prenatal ultrasound exam

SUMMARY:
Neural tube defects are one of the most prevalent congenital abnormalities, surpassed only by cardiac malformations. Spina bifida accounts for the majority of the neural tube defects and is comprised of a wide spectrum of anomalies ranging from small isolated sacral dysraphisms to large spinal defects. The origin of spina bifida is a failure of neurulation. It usually occurs at 15 days post-conception, resulting in a bony spinal defect with extrusion of the neural placode and/or the meninges outside of the spinal canal. Spina bifida has a prevalence of 1-5 in 1,000 live births and is the most complex congenital abnormality compatible to long-time survival. Concerning psychomotor development as well as urinary bladder and intestinal morbidity the prognosis ranges from normal functional outcome to severe disability.

The diagnosis of serious fetal abnormalities such as spinal dysraphism by ultrasound screening allows patients to prepare for the birth of an impaired child or to consider termination of the pregnancy. In current practice, prenatal counseling and obstetric management depend not only on the detection of a spinal dysraphism but also on an appropriate assessment of the severity of the defect and its possible impact on the postnatal development of the affected child.

Level and type of lesion, presence of associated anomalies (e.g., Chiari II malformation and ventriculomegaly) and mode of surgical closure are factors known to have prognostic impact on the postnatal outcome. Previous studies reported that postnatally determined lesion levels correlated well with functional status and survival. On the contrary, it is still not clear whether similar data obtained antenatally are of value.

In this study, the investigators will review their database of all cases of prenatally diagnosed spina bifida within a 16 year period between 1993 and 2009. By analyzing the prenatal and postnatal characteristics of fetuses with spina bifida in relation to the anatomic level of the lesion, the investigators aim to contribute further information regarding the natural course of affected pregnancies and the correlation of prenatal ultrasound findings with their functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* spina bifida identified at prenatal ultrasound examination
* ultrasound diagnosis between 1993 - 2009

Exclusion Criteria:

* deviant postnatal diagnosis
* loss to follow-up
* incomplete data

Ages: 12 Weeks to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fetuses with spina bifida identified at prenatal ultrasound examination between 1993 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2009-12; Primary Completion 2014-10 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
pregnancy outcome | 17 yrs
  To investigate the prenatal course and functional outcome of fetuses with spina bifida according to prenatal ultrasound exam.
Infant psychomotor development | 17 yrs
  Kaufmann ABC
  Denver Developmental Screening Test
  walking ability
  muscle strenght
Infant bladder and bowel function | 17 yrs
  Degree of continence.

SECONDARY OUTCOMES:
Conception date | 17 yrs
spectrum of ultrasound signs | 17yrs

CONTACTS AND LOCATIONS:
Overall Officials: Feriel Amari, M.D., Principal Investigator — Schleswig- Holstein University, Lübeck; Jan Weichert, M.D., Study Director — Schleswig- Holstein University, Lübeck; Klaus Diedrich, PhD, Study Chair — Schleswig- Holstein University, Lübeck
Locations (1):
- Schleswig- Holstein University, Campus Lübeck, Department of Prenatal Medicine, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Cameron M, Moran P. Prenatal screening and diagnosis of neural tube defects. Prenat Diagn. 2009 Apr;29(4):402-11. doi: 10.1002/pd.2250. PMID 19301349
- [Background] D'Addario V, Rossi AC, Pinto V, Pintucci A, Di Cagno L. Comparison of six sonographic signs in the prenatal diagnosis of spina bifida. J Perinat Med. 2008;36(4):330-4. doi: 10.1515/JPM.2008.052. PMID 18598123
- [Background] Biggio JR Jr, Owen J, Wenstrom KD, Oakes WJ. Can prenatal ultrasound findings predict ambulatory status in fetuses with open spina bifida? Am J Obstet Gynecol. 2001 Nov;185(5):1016-20. doi: 10.1067/mob.2001.117676. PMID 11717624
- [Background] Peralta CF, Bunduki V, Plese JP, Figueiredo EG, Miguelez J, Zugaib M. Association between prenatal sonographic findings and post-natal outcomes in 30 cases of isolated spina bifida aperta. Prenat Diagn. 2003 Apr;23(4):311-4. doi: 10.1002/pd.584. PMID 12673636
- [Derived] Beyer DA, Diedrich K, Weichert J, Kavallaris A, Amari F. Seasonality of spina bifida in Northern Germany. Arch Gynecol Obstet. 2011 Oct;284(4):849-54. doi: 10.1007/s00404-010-1762-0. Epub 2010 Nov 16. PMID 21079979